CLINICAL TRIAL: NCT02779426
Title: Texting Atopic Dermatitis Patients to Optimize Learning and EASI Scores
Acronym: TADPOLES
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Columbia University (Other)
Responsible Party: Principal Investigator, Christine Lauren, Assistant Professor of Dermatology and Pediatrics, Columbia University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: AAAQ7858
Record Dates: First submitted 2016-05-18; First posted 2016-05-20 (Estimated); Last update posted 2017-08-22 (Actual); Status verified 2017-08

CONDITIONS: Atopic Dermatitis
Keywords: Atopic dermatitis; Text Messages; Health literacy
MeSH Terms: conditions — Dermatitis, Atopic

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Text Message Intervention + Standard Care (Experimental): Enrolled patients and their caregivers who are randomized to this group will receive the usual standard of care for atopic dermatitis patients treated at this institution as well as daily text messages with information about atopic dermatitis and treatment reminders. 1-2 times/week they will receive a message asking if they were able to complete their treatments in the last day. They will respond with 1=yes, 2=no, 3= I have questions about the treatment. Those who respond with 3 will be sent the contact information for the office. No other communications will be sent through text messages. Caregivers will take two in-office surveys: one upon enrollment, and one follow-up survey at the follow-up visit. Patient EASI Score will be assessed by the pediatric dermatologist and initial and follow up exam.
  Interventions: Behavioral: Text messages
- Standard Care (No Intervention): Enrolled patients and their caregivers who are randomized to this group will receive the usual standard of care for atopic dermatitis patients treated at this institution. They will not receive text messages. Caregivers will take two in-office surveys: one upon enrollment, and one follow-up survey at the follow-up visit. Patient EASI Score will be assessed by the pediatric dermatologist and initial and follow up exam.

INTERVENTIONS:
Behavioral: Text messages — Daily text messages with information about atopic dermatitis and treatment reminders.
  Arms: Text Message Intervention + Standard Care

SUMMARY:
The purpose of this study is to determine if sending text messages with treatment reminders and facts regarding atopic dermatitis (AD) to caretakers of children with AD will have a positive effect on the disease severity.

DETAILED DESCRIPTION:
Atopic dermatitis (AD) is a common, chronic, and debilitating disease that tends to present in children under age 2 and has a waxing and waning course. Poor adherence to treatment is the primary preventable contributor towards adverse outcomes such as infection, hospitalization, permanent disfigurement, and disruptions in normal childhood psychological development. The burden of care for these patients often falls upon parents, who may have difficulty incorporating the necessary daily treatments into the family's lifestyle. Thus, investigating ways of improving adherence could have a significant impact on a patient's long term prognosis and the family's ability to understand and adjust to the demands of AD.Text message reminders with embedded health literacy information have been shown to improve vaccination rates in children and caregivers have reported increased satisfaction with this means of communication.

This study aims to assess whether text message reminders with information about AD are an effective way to improve treatment adherence and provide disease specific information to caregivers of children with AD. The measure of AD severity will be the Eczema Area and Severity Index (EASI) score. Health literacy with regard to AD will be assessed via in-office survey.This study will involve children age 0-6 with newly diagnosed AD and their primary caregivers. The subjects will be randomized to standard care or text message reminder group. All study participants will be asked to complete a survey after their initial evaluation and after their follow up visit on the same day they are in the office. The text message group will receive text messages with information and treatment reminders. All participants will receive the standard of care with regard to AD.

If this study demonstrates that text message reminders can improve EASI scores in AD patients it could lead to a significant change in how these patients are managed. Fewer complications from episodic flares, infections, and other sequelae may lessen the burden of this disease for both patients and their caregivers. Text messaging is an inexpensive, noninvasive, and broadly applicable tool that is worth studying for the purpose of improving treatment adherence and disease literacy.

ELIGIBILITY:
Inclusion Criteria:

* New clinical diagnosis of atopic dermatitis
* New patient to Columbia University Medical Center, Department of Dermatology
* Caregiver has mobile that can send/receive text messages

Exclusion Criteria:

* Age over 7 years
* Caregiver is not fluent English speaker
* Those patients in which a definitive diagnosis of atopic dermatitis cannot be made
* Any individual who declines participation

Max Age: 6 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 84 (Actual)
Dates: Start 2016-05 (Actual); Primary Completion 2017-06 (Actual); Study Completion 2017-07 (Actual)

PRIMARY OUTCOMES:
EASI Score | Up to 6 weeks
  Patient EASI Score (0-72) will be determined at initial and follow up exam. Mean differences in EASI scores between arms will be assessed using t-tests since EASI scores are used to measure the severity of a patient's atopic dermatitis.

SECONDARY OUTCOMES:
Patient Satisfaction | Up to 6 weeks
  The investigators will assess mean difference in reported satisfaction, as indicated on follow up survey, between arms using t-tests.

CONTACTS AND LOCATIONS:
Overall Officials: Christine Lauren, MD, Principal Investigator — Columbia University
Locations (1):
- Columbia University Medical Center, Department of Dermatology, New York, New York, United States

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Sokolova A, Smith SD. Factors contributing to poor treatment outcomes in childhood atopic dermatitis. Australas J Dermatol. 2015 Nov;56(4):252-7. doi: 10.1111/ajd.12331. Epub 2015 Mar 29. PMID 25817780
- [Background] Filanovsky MG, Pootongkam S, Tamburro JE, Smith MC, Ganocy SJ, Nedorost ST. The Financial and Emotional Impact of Atopic Dermatitis on Children and Their Families. J Pediatr. 2016 Feb;169:284-90.e5. doi: 10.1016/j.jpeds.2015.10.077. Epub 2015 Nov 23. PMID 26616249
- [Background] Bass AM, Anderson KL, Feldman SR. Interventions to Increase Treatment Adherence in Pediatric Atopic Dermatitis: A Systematic Review. J Clin Med. 2015 Jan 27;4(2):231-42. doi: 10.3390/jcm4020231. PMID 26239125
- [Background] Stockwell MS, Hofstetter AM, DuRivage N, Barrett A, Fernandez N, Vargas CY, Camargo S. Text message reminders for second dose of influenza vaccine: a randomized controlled trial. Pediatrics. 2015 Jan;135(1):e83-91. doi: 10.1542/peds.2014-2475. PMID 25548329